CLINICAL TRIAL: NCT07196891
Title: Prognostic Value of the Frontal QRS/T Angle for 28-day Mortality and Neurological Outcomes in Aneurysmal Subarachnoid Hemorrhage
Brief Title: Predictive Role of f-QRST Angle in Subarachnoid Hemorrhage
Acronym: f-QRST in SAH
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: 135-2025
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Subarachnoid Hemorrhage; Aneurysmal; Non-traumatic; Electrocardiography; frontal-QRST angle; 28-day mortality
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Survivors were defined as patients who were still alive after 28 days of admission to the emergency department.
  Interventions: Other: frontal-QRST angle; Other: Hunt-Hess scale; Other: modified Fisher scale
- Non-survivors: Non-survivors had passed away within 28 days of admission to the emergency department.
  Interventions: Other: frontal-QRST angle; Other: Hunt-Hess scale; Other: modified Fisher scale

INTERVENTIONS:
Other: frontal-QRST angle — The frontal QRS/T angle represents the angle between the ventricular depolarization (QRS) and repolarization (T) vectors on the ECG and serves as a parameter for assessing cardiac electrical heterogeneity. In this study, the frontal QRS/T angle was calculated using data obtained from standard 12-lead surface ECGs. The QRS and T axes in the frontal plane were derived from the automated ECG device reports.
Other: Hunt-Hess scale — The Hunt-Hess scale was used to assess SAH severity according to the clinical presentation and the visible neurological deficits. The Grades run from 1 to 5: - Grade 1: Asymptomatic or minimal headache, slight neck stiffness. - Grade 2: Moderate to severe headache, and neck stiffness, but no neurological deficit except cranial nerve palsy. - Grade 3: Drowsiness, confusion, or a mild focal deficit. - Grade 4: Stupor, moderate to severe hemiparesis, early decerebrate rigidity, and vegetative disturbance. - Grade 5: Deep coma, decerebrate rigidity, and a moribund appearance.
Other: modified Fisher scale — The modified Fisher scale was used to evaluate SAH severity by reference to the extent of hemorrhage as revealed by CT of the brain. Four grades are depending on the degree of bleeding observed: - Grade 0: No hemorrhage apparent in CT. - Grade 1: Minimal hemorrhage without intraventricular hemorrhage (IVH). - Grade 2: Thin or diffusely thin (<1mm) hemorrhage with bilateral IVH. - Grade 3: Thick (> 1 mm) hemorrhage without bilateral IVH. - Grade 4: Thick (> 1 mm) hemorrhage with bilateral IVH.

SUMMARY:
The investigators investigated the association between the frontal QRS/T angle measured on admission ECG and 28-day mortality, as well as neurological outcome in patients with non-traumatic aneurysmal SAH. Specifically, the investigators tested the hypothesis that an increased frontal QRS/T angle would be independently associated with higher mortality and poorer clinical outcomes in patients with SAH. Accordingly, the investigators also analyzed the relationship between the frontal QRS/T angle and neurological status assessed based on Glasgow Outcome Scale (GOS), as well as disease severity determined by the Hunt-Hess and Fisher grading systems.

DETAILED DESCRIPTION:
Patients were divided into two groups: survivors and non-survivors. Survivors were further classified as mobile or immobile according to the Glasgow Outcome Scale (GOS). Patients who remained comatose or dependent in daily activities were classified as immobile (GOS 1-3), while those who returned to normal life or were able to perform daily activities independently were classified as mobile (GOS 4-5). Demographic and clinical characteristics as well as ECG findings were compared between these groups, and the relationship between the frontal QRS/T angle, 28-day mortality, and disease severity was evaluated. Independent predictors of mortality were determined by multivariate logistic regression analysis of variables (demographic characteristics, clinical characteristics, and ECG changes) that differed significantly between survivors and non-survivors. An area under the curve (AUC) analysis was then conducted to identify the predictive role of the f-QRST angle in patients with SAH.

ELIGIBILITY:
Inclusion Criteria:

- patients (aged ≥ 18 years) who presented to the emergency department with non-traumatic Subarachnoid Hemorrhage between July 2020 and July 2025

Exclusion Criteria:

* patients younger than 18 years
* patients with missing information
* patients with traumatic SAH
* patients with subdural or epidural hemorrhage
* patients with concurrent ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter, retrospective, observational cohort study enrolled 354 consecutive adult patients (aged ≥ 18 years) who presented to the emergency departments of the seven major and highest-volume tertiary hospitals in Istanbul with non-traumatic Subarachnoid Hemorrhage between July 2020 and July 2025. Data were collected by searching for I60.9 International Classification of Diseases (ICD) codes in the hospital's automation systems and archives.
Sampling Method: Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Predictive ability of frontal-QRST angle for 28-day mortality | From admission to 28 days
  The investigators assessed the predictive ability of frontal-QRST angle in determining 28-day mortality.

SECONDARY OUTCOMES:
Predictive ability of frontal-QRST angle for neurological survival | From admission to 28 days
  The investigators assessed the predictive ability of frontal-QRST angle in determining neurological survival

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Background] Gunduz R, Yildiz BS, Ozgur S, Ozen MB, Bakir EO, Ozdemir IH, Cetin N, Usalp S, Duman S. Frontal QRS/T angle can predict mortality in COVID-19 patients. Am J Emerg Med. 2022 Aug;58:66-72. doi: 10.1016/j.ajem.2022.05.034. Epub 2022 May 25. PMID 35636045
- [Background] Hocanli I, Tanriverdi Z, Kabak M, Gungoren F, Tascanov MB. The relationship between frontal QRS-T angle and the severity of newly diagnosed chronic obstructive pulmonary disease. Int J Clin Pract. 2021 Oct;75(10):e14500. doi: 10.1111/ijcp.14500. Epub 2021 Jun 29. PMID 34117683
- [Background] Zhang X, Zhu Q, Zhu L, Jiang H, Xie J, Huang W, Xu B. Spatial/Frontal QRS-T Angle Predicts All-Cause Mortality and Cardiac Mortality: A Meta-Analysis. PLoS One. 2015 Aug 18;10(8):e0136174. doi: 10.1371/journal.pone.0136174. eCollection 2015. PMID 26284799
- [Background] Bilginer HA, Sogut O, Az A, Ergenc H. Electrocardiographic abnormalities are prognostic of the clinical outcomes and mortality of patients with subarachnoid hemorrhages. Am J Emerg Med. 2024 Jul;81:140-145. doi: 10.1016/j.ajem.2024.04.055. Epub 2024 May 3. PMID 38728937
- [Background] Thilak S, Brown P, Whitehouse T, Gautam N, Lawrence E, Ahmed Z, Veenith T. Diagnosis and management of subarachnoid haemorrhage. Nat Commun. 2024 Feb 29;15(1):1850. doi: 10.1038/s41467-024-46015-2. PMID 38424037
- [Background] Cetinkaya O, Arslan U, Temel H, Kavakli AS, Cakin H, Cengiz M, Yilmaz M, Barcin NE, Ikiz F. Factors Influencing the Mortality of Patients with Subarachnoid Haemorrhage in the Intensive Care Unit: A Retrospective Cohort Study. J Clin Med. 2025 Feb 28;14(5):1650. doi: 10.3390/jcm14051650. PMID 40095649